CLINICAL TRIAL: NCT01021189
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD1446 in Healthy Young and Elderly Japanese Volunteers After Oral Single and Multiple Ascending Doses
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics After Single and Multiple Doses of AZD1446 to Japanese Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1950C00003
Record Dates: First submitted 2009-11-23; First posted 2009-11-26 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: safety; tolerability; AZD1446; AD; Japanese
MeSH Terms: interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD1446
  Interventions: Drug: AZD1446
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1446 — Oral solution Dose single and followed by 7-day multiple dosing.Specific doses depend on panel.
  Arms: 1
Drug: Placebo — Oral solution Dose single and followed by 7-day multiple dosing.
  Arms: 2

SUMMARY:
The primary aim of this study is to assess the safety and tolerability of AZD1446 following single and multiple ascending doses of an orally administered solution of AZD1446 in healthy young and elderly Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese subjects, aged ≥20 to ≤50 years for male young subjects, ≥65 to ≤80 years for male or post-menopausal female elderly subjects.
* BMI between 18 and 27 kg/m2 and weigh at least 50 kg and no more than 90 kg (for the elderly female, weigh at least 45 kg and no more than 90 kg).

Exclusion Criteria:

* History of Quincke oedema or angiooedema, or history of repeated episodes of urticaria.
* History or present symptoms or signs of asthma, airway hyperreactivity or obstructive lung disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD1446 following single and multiple ascending doses of an orally administered solution of AZD1446 in healthy young and elderly Japanese subjects by adverse events, vital signs, laboratory variables and ECG. | During the whole study period, ca. 50 days.

SECONDARY OUTCOMES:
To determine pharmacokinetics(PK) of AZD1446 following single and multiple dosing of AZD1446 in healthy young and elderly Japanese subjects. | PK sampling taken at defined timepoints during residential period, 12 days.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Paulsson, MD, PhD, Study Director — AstraZeneca R&D Södertälje; Shunji Matsuki, MD, PhD, Principal Investigator — Kyusyu Clinical Phramacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Japan